CLINICAL TRIAL: NCT02590692
Title: A Phase I/IIa Safety Study of Subretinal Implantation of CPCB-RPE1 (Human Embryonic Stem Cell-Derived Retinal Pigment Epithelial Cells Seeded on a Polymeric Substrate) in Subjects With Advanced, Dry Age-Related Macular Degeneration (AMD)
Brief Title: Study of Subretinal Implantation of Human Embryonic Stem Cell-Derived RPE Cells in Advanced Dry AMD
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Regenerative Patch Technologies, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RPT-14-01
Record Dates: First submitted 2015-10-23; First posted 2015-10-29 (Estimated); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Dry Macular Degeneration; Geographic Atrophy
MeSH Terms: conditions — Geographic Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CPCB-RPE1 treatment (Experimental): Subretinal implantation of CPCB-RPE1 in dry AMD patients
  Interventions: Biological: CPCB-RPE1

INTERVENTIONS:
Biological: CPCB-RPE1 — Patients will receive one CPCB-RPE1 implant of approximately 100,000 differentiated RPE cells attached to a small parylene membrane. The density of cells on the membrane represents the approximate density of RPE cells in the human eye. The membrane size was chosen to cover a substantial portion of the macular region of the retina.

SUMMARY:
The Phase I/IIa clinical trial is designed to assess the feasibility of delivery and safety of Human Embryonic Stem Cell-Derived RPE Cells on a parylene membrane (CPCB-RPE1) in patients with advanced, dry age-related macular degeneration.

Primary Objective:

• To test the safety and tolerability of CPCB-RPE1 during and after subretinal implantation in patients with geographic atrophy with evidence of involvement of the central fovea.

Secondary Objective:

• To assess visual acuity, visual field, and retinal function after CPCB-RPE1 implantation. Implanted and fellow eyes will be compared post-implantation to assess the ability of the implant to prevent disease progression.

Exploratory Objectives:

• To assess the feasibility of measuring the change in area of geographic atrophy over time using spectral domain optical coherence tomography or fundus autofluorescence.

DETAILED DESCRIPTION:
The study will include two cohorts, each of 10 patients. For the first cohort, the study population will be patients with advanced, dry AMD with evidence of significant geographic atrophy involving the fovea. These patients will have significant central vision loss with best-corrected visual acuity (BCVA) of the eye to be implanted of BCVA of 20/200 or worse. Each of these patients will have substantial RPE and photoreceptor loss. Patients will be screened for overall health status to minimize risks associated with retinal surgery and any subsequent immunosuppression.

As the safety and tolerability of CPCB-RPE1 is demonstrated in the first cohort, patients with less advanced disease will be recruited into a second cohort in this Phase I/IIa clinical trial. In this second cohort patients will have significant central vision loss with BCVA of the eye to be implanted of 20/80 or worse, but better than or equal to 20/400 with comparably less damage to the RPE/photoreceptor complex than Cohort 1. These patients will be screened in the same manner for overall health status to minimize risks associated with retinal surgery and any subsequent immunosuppression. Assessments of visual function will be the same as in Cohort 1.

ELIGIBILITY:
Inclusion Criteria:

1. Patients able to understand and willing to sign the informed consent
2. Adult male or female patients with the age of 55 to 85 (inclusive) years who are not employees of the trial sites
3. In sufficiently good health to reasonably expect survival for at least five years after treatment
4. Clinical findings consistent with advanced dry AMD with evidence of one or more areas of ≥1.25 square millimeter of geographic atrophy involving the central fovea
5. Geographic atrophy defined as attenuation or loss of RPE as observed by biomicroscopy, OCT, or FAF
6. The best-corrected visual acuity (BCVA) of the eye to receive the implant will be equal or worse than 20/200 in the first half of the study patients and between 20/80 and 20/400 (inclusive) in the second half of the patients. The BCVA of the eye that is NOT to receive the implant will be better or equal to the eye that will receive the implant
7. Medically suitable to undergo pars plana vitrectomy and the surgical implant procedure, including being able to position post-operatively and use post-operative medications as required
8. Medically suitable for general anesthesia or monitored intravenous sedation, if needed
9. Patients who are pseudophakic or aphakic in the study eye
10. If designated as an organ donor, willing to forego live organ donation
11. Willing to consent to the post-mortem removal of the implant from the treated eye for the sponsor's analysis. The patient may also elect to donate the implanted and fellow, untreated eye, for histological analysis.
12. Able to understand the requirements of the study and willing and able to participate in long term follow up.

Exclusion Criteria:

1. Presence of active or inactive choroidal neovascularization (CNV)
2. Presence or history of retinal dystrophy, retinitis pigmentosa, chorioretinitis, central serous choroidopathy or any other inflammatory ocular disease except dry eye syndrome
3. Presence or history of severe, end-stage corneal dystrophy
4. History of steroid induced ocular hypertension or glaucoma
5. Presence of moderate to severe glaucomatous optic neuropathy in the study eye, uncontrolled IOP, use of two or more topical agents to control intraocular pressure; history of glaucoma-filtering surgery
6. Presence of moderate to severe non-proliferative diabetic retinopathy in the study eye
7. Presence of any proliferative diabetic retinopathy in the study eye
8. Presence of uncontrolled diabetes mellitus (HbA1c > 8) at the time of screening
9. History of retinal detachment or retinal detachment repair in the study eye other than peripheral retinal tears or holes treated exclusively with laser or cryotherapy
10. Presence of any other sight-threatening ocular disease
11. History of cognitive impairments or dementia which may impact the patient's ability to participate in the informed consent process and to appropriately complete evaluations
12. History of any immunodeficiency
13. Evidence of herpetic or other viral eye disease
14. Any current use of immunosuppressive therapy other than intermittent or low dose corticosteroids
15. Participation within previous 3 months in any clinical trial of a drug by ocular or systemic administration (within previous 18 months for sustained release products)
16. Axial myopia of greater than -8 diopters in the eye that is to be implanted
17. Axial length greater than 28 mm in the eye that is to be implanted
18. History of malignancy within the past 5 years (with the exception of successfully treated [excised] basal cell carcinoma [skin cancer] or successfully treated squamous cell carcinoma of the skin)
19. History of myocardial infarction in previous 12 months
20. Alanine transaminase/aspartate aminotransferase (ALT/AST) >3.0 times the upper limit of normal or any known liver disease
21. Renal insufficiency, as defined by estimated creatinine clearance of < 45 ml/min
22. A positive (or "reactive") test for HIV, or Hepatitis B, or Hepatitis C
23. A hemoglobin concentration of less than 10 gm/dl, a platelet count of less than 100K/µL or an absolute neutrophil count of less than 1000/µL at study entry
24. Ocular lens removal within the previous 6 weeks in either eye
25. Any other ocular surgery in the study eye in the previous 3 months
26. If female, pregnancy, the wish to become pregnant, or lactation
27. Any other medical condition, which, in the Investigator's judgment, will interfere with the patient's ability to comply with the protocol, compromises patient safety, or interferes with the interpretation of the study results

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-02-16 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Frequency and Severity of Treatment-Related Adverse Events [Safety and Tolerability] | 1 year
  Comparison of product, procedure and immunosuppression related adverse events in the implanted eye to those experienced in the non-treated eye

SECONDARY OUTCOMES:
Visual Acuity | 1 year
  Comparison of VA changes in the treated eye versus baseline and versus the non-treated eye
Visual Field | 1 year
  Comparison of visual field changes in the treated eye versus baseline and versus the non-treated eye
Photoreceptor Electrical Responses | 1 year
  Comparison of multifocal electroretinogram changes in the treated eye versus baseline and versus the non-treated eye

CONTACTS AND LOCATIONS:
Overall Officials: Jane Lebkowski, Ph.D., Study Director — Regenerative Patch Technologies
Locations (6):
- United States (6):
  - Retinal Consultants of Arizona LTD, Phoenix, Arizona
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - USC Keck School of Medicine / Eye Institute, Los Angeles, California
  - Southern California Desert Retina Consultants, Palm Desert, California
  - Orange County Retina Medical Group, Santa Ana, California
  - California Retina Consultants, Santa Barbara, California